CLINICAL TRIAL: NCT01946997
Title: Evaluation of the Retina of Subjects Without Diabetes Mellitus and Subjects With Diabetes Mellitus Without Diabetic Retinopathy Using Optical Coherence Tomography
Status: Completed | Type: Observational
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Other Study IDs: 03-11-05-03
Record Dates: First submitted 2013-09-17; First posted 2013-09-20 (Estimated); Last update posted 2017-12-06 (Actual); Status verified 2017-12

CONDITIONS: Diabetic Retinopathy
MeSH Terms: conditions — Diabetic Retinopathy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group 1: Non Diabetic: Normal retina
  Interventions: Other: OCT Imaging both Normal and diabetic groups
- Group 2: Diabetes with no retinopathy: Diabetic patients without diabetic retinopathy
  Interventions: Other: OCT Imaging both Normal and diabetic groups

INTERVENTIONS:
Other: OCT Imaging both Normal and diabetic groups — Images taken to determine thickness values in the retina
  Other Names: Ocular Coherence tomography

SUMMARY:
The purpose of this study is to evaluate topographic features of the posterior pole of the eye in normal subjects as well as in subjects with diabetes mellitus but without diabetic retinopathy (DR) using optical coherence tomography (OCT). The investigators proposal is a novel study to determine retinal volume of normal and diabetic subjects without DR. Specifically, the investigators will establish a standardized reference range for retinal thickness and volume that will provide standards for OCT analysis of different clinical trials for retinal diseases.

ELIGIBILITY:
Inclusion Criteria:

* Healthy retinas
* Willingness to sign informed consent to have OCT images taken.

Exclusion Criteria:

* No macular pathology
* No Diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Normal, non-diabetic patients
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2006-07; Primary Completion 2009-11 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Normative retinal thickness data for comparison | one year
  Normative retinal thickness data for comparison

CONTACTS AND LOCATIONS:
Overall Officials: Quan D Nguyen, MD, MSc, Principal Investigator — Johns Hopkins University